CLINICAL TRIAL: NCT01495767
Title: The Impact of Uveitis on Health-related Quality of Life in Adolescents
Brief Title: Quality of Life in Juvenile Patients With Uveitis
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Saskia M Maca, MD, principal investigator, Hospital Hietzing
Other Study IDs: MAC205
Record Dates: First submitted 2011-11-27; First posted 2011-12-20 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Uveitis
Keywords: childhood uveitis; health-related quality of life; gender
MeSH Terms: conditions — Uveitis; Coitus

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- females, males: females: patients of female sex males: patients of male sex
  Interventions: Other: Filling in a psychometric questionnaire

INTERVENTIONS:
Other: Filling in a psychometric questionnaire — Juvenile patients attending the uveitis are asked to fill in a psychometric questionnaire

SUMMARY:
Data about psychodynamics in uveitis patients are scare. A negative impact of disease is described not only in adult patients with active, but also with quiescent disease. During adolescence even less is known about psychodynamics although this is an especially sensible and challenging stage of life. Given the assumption that juvenile patients with quiescent disease still could suffer from emotional distress, this would require special attention.

In this study the investigators evaluate the impact of juvenile uveitis on HRQoL and attempted to identify clinical and demographic factors contributing to an impaired health status. The investigators limit the study to patients with quiescent uveitis and good visual function in at least one eye to exclude additional negative stressors. As there are no validated uveitis-specific psychometric questionnaires evaluating QoL available yet, the investigators use age-appropriate generic instruments. This should allow obtaining an overview about the adolescents' general Health-related Quality of Life (HRQoL) and whether psychological interventions should be offered to this sensitive patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with uveitis
* aged 11-18 years
* willing to participate
* parent or legal guardian agrees with participation of adolescent

Exclusion Criteria:

* not willing to participate
* parent or legal guardian does not agree with participation of adolescent

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with uveitis, aged 11-18 years
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2006-01; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Quality of life as assessed with the "Inventory for Assessing the Quality of Life in Children and Adolescents" | One day
  psychometric inventory

SECONDARY OUTCOMES:
Quality of life as assessed with the "Children Quality of Life Questionnaire" | One day
  psychometric inventory

CONTACTS AND LOCATIONS:
Overall Officials: Saskia M Maca, MD, Principal Investigator — Hospital Hietzing, Vienna + Medical University of Vienna, Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria